CLINICAL TRIAL: NCT02956096
Title: Evaluation of Autonomic Modulation in the Hemiparetic Patients After Transcranial Direct Current Stimulation (tDCS) and Treadmill Training: Clinical Trial, Controlled, a Randomized, Double-blind
Brief Title: Evaluation of Autonomic Modulation in Stroke After Transcranial Direct Current Stimulation and Treadmill Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Glauber Heinz, Physiotherapist, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: u64963ep
Record Dates: First submitted 2016-09-30; First posted 2016-11-04 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: tDCS; Stroke; Autonomic Modulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tDCS device and Treatmill (Active Comparator): The stimulation is accomplished with a direct current-tDCS Stimulator Plus device, via two surface electrodes sponge (non-metallic) 5-7 cm2 in saline moistened with a 2mA current during 20 minutes after hemodinamic analysis is performed for 15 minutes and then made only training treadmill for 20 minutes. Placebo tDCS will follow the same procedures, but the tDCS device will only be switched on for 20 seconds. The running in the treadmill will be held on a single training session and the speed of the cardiopulmonary exercise testing and slope from 60 to 80% of the maximum achieved in cardiopulmonary testing, in order that the patient reaches 60% to 70% of the heart rate reserve (MACKO , 2005).
  Interventions: Device: Transcranial direct current stimulation (tDCS); Device: training on the running belt
- 1- tDCS (Sham Comparator): 1. Who received stimulation transcranial direct current active will receive Sham stimulation and who received the placebo stimulation receive active stimulation and then the two groups will do the workout on the treadmill
  Interventions: Device: Transcranial direct current stimulation (tDCS); Device: training on the running belt

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — The active tDCS and placebo will be applied to anode electrode on left temporal cortex placed on the scalp in the region T3. The cathode electrode on the middle deltoid muscle contralateral to the anode.
Device: training on the running belt — The running in the treadmill will be held on a single training session and the speed of the cardiopulmonary exercise testing and slope from 60 to 80% of the maximum achieved in cardiopulmonary testing, in order that the patient reaches 60% to 70% of the heart rate reserve.

SUMMARY:
Introduction: Patients post-stroke may have autonomic dysfunction, with increased blood pressure, heart rate (HR) and increased risk of sudden death. Studies have shown that transcranial direct-current stimulation (tDCS) can modulate the autonomic nervous system in healthy subjects, but little is known about these effects in stroke.

Objective: To evaluate the effect of tDCS after treadmill training in the autonomic nervous system modulation in patients post-stroke.

DETAILED DESCRIPTION:
Introduction: Patients post-stroke may have autonomic dysfunction, with increased blood pressure, heart rate (HR) and increased risk of sudden death. Studies have shown that transcranial direct-current stimulation (tDCS) can modulate the autonomic nervous system in healthy subjects, but little is known about these effects in stroke.

Objective: To evaluate the effect of tDCS after treadmill training in the autonomic nervous system modulation in patients post-stroke.

Methods: Clinical study, crossover, controlled, randomized, double-blind individuals with hemiparesis after stroke adults. Patients will undergo a spirometric evaluation (Harbor protocol modified with constant speed, determined by the individual and the incline of the treadmill with incremented 2.5% every 2 minutes). The next day will begin with one of the two randomized protocols, one week interval between them: 1 (tDCS active and treadmill), 2 (tDCS placebo and treadmill). Each protocol will last 40 minutes (20min of tDCS over 20min mat). They will be evaluated heart rate variability (HRV) and blood pressure variability (VPA) before a minute for the protocols and in the recovery phase, for 15 minutes. 2mA current intensity, the anode electrode over the left temporal cortex and cathode on the contralateral deltoid muscle. Considering the neurophysiological effects of noninvasive techniques neuromodulators plasticity before the modulation of the autonomic nervous system, it is concluded that this study shows potential for the discovery of a new therapeutic tool in the rehabilitation of patients with stroke and hypertension. The hypothesis is that increasing the excitability of the left insular cortex, a modulation of the autonomic nervous system in controlling the variability in systolic blood pressure and heart rate is possible in conjunction with aerobic training, can provide greater hemodynamic effectiveness and decrease the time training. It is also understood that the study may have impact on the reduction of public costs spent on the rehabilitation of patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* present hemiparesis due to stroke for more than 6 months;
* Commitment mild or moderate motor in the lower member (20 to 31 points), according to the scores of Fugl-Meyer test
* comfortable walking speed on the ground between 0.3 and 1.15 m / s;
* Rating between levels 04-06 on Functional Mobility Scale (FMS) - Functional Mobility Scale and ambulate at least 50 meters
* Presentation of the AVE imaging
* Science Signature regarding the free and informed consent (WIC).

Exclusion Criteria:

* present cognitive impairment (mini mental) with scores below 24 points;
* visual impairment that may interfere with the performance of the tests;
* severe heart failure (congestive heart failure, angina, peripheral vascular disease), pacemaker use, β-blockers and propranolol;
* contraindications to the use of tDCS (brain implants of metal clips near the region to be stimulated, history of recurrent seizures, recurrent epilepsy and brain tumors, brain pacemaker and / or plates or metal devices in place of stimulation tDCS)
* irregular menstrual cycle or be in the menstrual period during the evaluation;
* No medical certificate for treadmill exercise test

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 1 years
  Cardiac Frequency Variability (HRV) as measured by spectral analysis by Finomiter (FMS, Finapres Measurement Systems, Arnhem, Netherlands), in ms²

SECONDARY OUTCOMES:
Blood pressure variability | 1 years
  Blood Pressure Variability (BPV) as measured by spectral analysis by Finomiter (FMS, Finapres Measurement Systems, Arnhem, Netherlands), in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- University Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Qudah ZA, Yacoub HA, Souayah N. Disorders of the Autonomic Nervous System after Hemispheric Cerebrovascular Disorders: An Update. J Vasc Interv Neurol. 2015 Oct;8(4):43-52. PMID 26576215
- [Background] Verberne AJ, Owens NC. Cortical modulation of the cardiovascular system. Prog Neurobiol. 1998 Feb;54(2):149-68. doi: 10.1016/s0301-0082(97)00056-7. PMID 9481796
- [Background] Billinger SA, Arena R, Bernhardt J, Eng JJ, Franklin BA, Johnson CM, MacKay-Lyons M, Macko RF, Mead GE, Roth EJ, Shaughnessy M, Tang A; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Epidemiology and Prevention; Council on Clinical Cardiology. Physical activity and exercise recommendations for stroke survivors: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Aug;45(8):2532-53. doi: 10.1161/STR.0000000000000022. Epub 2014 May 20. PMID 24846875
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Christensen H, Boysen G, Christensen AF, Johannesen HH. Insular lesions, ECG abnormalities, and outcome in acute stroke. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):269-71. doi: 10.1136/jnnp.2004.037531. PMID 15654050
- [Background] Colivicchi F, Bassi A, Santini M, Caltagirone C. Prognostic implications of right-sided insular damage, cardiac autonomic derangement, and arrhythmias after acute ischemic stroke. Stroke. 2005 Aug;36(8):1710-5. doi: 10.1161/01.STR.0000173400.19346.bd. Epub 2005 Jul 14. PMID 16020766
- [Background] Eckardt M, Gerlach L, Welter FL. Prolongation of the frequency-corrected QT dispersion following cerebral strokes with involvement of the insula of Reil. Eur Neurol. 1999;42(4):190-3. doi: 10.1159/000008105. PMID 10567813
- [Background] Graham HK, Harvey A, Rodda J, Nattrass GR, Pirpiris M. The Functional Mobility Scale (FMS). J Pediatr Orthop. 2004 Sep-Oct;24(5):514-20. doi: 10.1097/00004694-200409000-00011. PMID 15308901
- [Background] Kang J, Hong JH, Jang MU, Kim BJ, Bae HJ, Han MK. Cardioembolism and Involvement of the Insular Cortex in Patients with Ischemic Stroke. PLoS One. 2015 Oct 21;10(10):e0139540. doi: 10.1371/journal.pone.0139540. eCollection 2015. PMID 26489090
- [Background] Kluding PM, Tseng BY, Billinger SA. Exercise and executive function in individuals with chronic stroke: a pilot study. J Neurol Phys Ther. 2011 Mar;35(1):11-7. doi: 10.1097/NPT.0b013e318208ee6c. PMID 21475079
- [Background] Macey PM, Wu P, Kumar R, Ogren JA, Richardson HL, Woo MA, Harper RM. Differential responses of the insular cortex gyri to autonomic challenges. Auton Neurosci. 2012 May 21;168(1-2):72-81. doi: 10.1016/j.autneu.2012.01.009. Epub 2012 Feb 17. PMID 22342370
- [Background] Macko RF, Ivey FM, Forrester LW, Hanley D, Sorkin JD, Katzel LI, Silver KH, Goldberg AP. Treadmill exercise rehabilitation improves ambulatory function and cardiovascular fitness in patients with chronic stroke: a randomized, controlled trial. Stroke. 2005 Oct;36(10):2206-11. doi: 10.1161/01.STR.0000181076.91805.89. Epub 2005 Sep 8. PMID 16151035
- [Background] Makovac E, Thayer JF, Ottaviani C. A meta-analysis of non-invasive brain stimulation and autonomic functioning: Implications for brain-heart pathways to cardiovascular disease. Neurosci Biobehav Rev. 2017 Mar;74(Pt B):330-341. doi: 10.1016/j.neubiorev.2016.05.001. Epub 2016 May 13. PMID 27185286
- [Background] Pang MY, Eng JJ, Dawson AS, Gylfadottir S. The use of aerobic exercise training in improving aerobic capacity in individuals with stroke: a meta-analysis. Clin Rehabil. 2006 Feb;20(2):97-111. doi: 10.1191/0269215506cr926oa. PMID 16541930
- [Background] Nagai M, Hoshide S, Kario K. The insular cortex and cardiovascular system: a new insight into the brain-heart axis. J Am Soc Hypertens. 2010 Jul-Aug;4(4):174-82. doi: 10.1016/j.jash.2010.05.001. PMID 20655502
- [Background] Noetscher GM, Yanamadala J, Makarov SN, Pascual-Leone A. Comparison of cephalic and extracephalic montages for transcranial direct current stimulation--a numerical study. IEEE Trans Biomed Eng. 2014 Sep;61(9):2488-98. doi: 10.1109/TBME.2014.2322774. PMID 25014947
- [Background] Oppenheimer SM, Gelb A, Girvin JP, Hachinski VC. Cardiovascular effects of human insular cortex stimulation. Neurology. 1992 Sep;42(9):1727-32. doi: 10.1212/wnl.42.9.1727. PMID 1513461
- [Background] Oppenheimer SM, Kedem G, Martin WM. Left-insular cortex lesions perturb cardiac autonomic tone in humans. Clin Auton Res. 1996 Jun;6(3):131-40. doi: 10.1007/BF02281899. PMID 8832121
- [Background] Lista Paz A, Gonzalez Doniz L, Ortigueira Garcia S, Saleta Canosa JL, Moreno Couto C. Respiratory Muscle Strength in Chronic Stroke Survivors and Its Relation With the 6-Minute Walk Test. Arch Phys Med Rehabil. 2016 Feb;97(2):266-72. doi: 10.1016/j.apmr.2015.10.089. Epub 2015 Oct 28. PMID 26519610
- [Background] Montenegro RA, Farinatti Pde T, Fontes EB, Soares PP, Cunha FA, Gurgel JL, Porto F, Cyrino ES, Okano AH. Transcranial direct current stimulation influences the cardiac autonomic nervous control. Neurosci Lett. 2011 Jun 15;497(1):32-6. doi: 10.1016/j.neulet.2011.04.019. Epub 2011 Apr 17. PMID 21527314
- [Background] Roth EJ. Heart disease in patients with stroke. Part II: Impact and implications for rehabilitation. Arch Phys Med Rehabil. 1994 Jan;75(1):94-101. PMID 8291971
- [Background] Ruggiero DA, Mraovitch S, Granata AR, Anwar M, Reis DJ. A role of insular cortex in cardiovascular function. J Comp Neurol. 1987 Mar 8;257(2):189-207. doi: 10.1002/cne.902570206. PMID 3571525
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Scheitz JF, Erdur H, Haeusler KG, Audebert HJ, Roser M, Laufs U, Endres M, Nolte CH. Insular cortex lesions, cardiac troponin, and detection of previously unknown atrial fibrillation in acute ischemic stroke: insights from the troponin elevation in acute ischemic stroke study. Stroke. 2015 May;46(5):1196-201. doi: 10.1161/STROKEAHA.115.008681. Epub 2015 Apr 2. PMID 25835563
- [Background] Smith AC, Saunders DH, Mead G. Cardiorespiratory fitness after stroke: a systematic review. Int J Stroke. 2012 Aug;7(6):499-510. doi: 10.1111/j.1747-4949.2012.00791.x. Epub 2012 May 9. PMID 22568786
- [Background] Soros P, Hachinski V. Cardiovascular and neurological causes of sudden death after ischaemic stroke. Lancet Neurol. 2012 Feb;11(2):179-88. doi: 10.1016/S1474-4422(11)70291-5. PMID 22265213
- [Background] De Raedt S, De Vos A, De Keyser J. Autonomic dysfunction in acute ischemic stroke: an underexplored therapeutic area? J Neurol Sci. 2015 Jan 15;348(1-2):24-34. doi: 10.1016/j.jns.2014.12.007. Epub 2014 Dec 8. PMID 25541326
- [Background] Tokgozoglu SL, Batur MK, Topcuoglu MA, Saribas O, Kes S, Oto A. Effects of stroke localization on cardiac autonomic balance and sudden death. Stroke. 1999 Jul;30(7):1307-11. doi: 10.1161/01.str.30.7.1307. PMID 10390300
- [Background] Triposkiadis F, Karayannis G, Giamouzis G, Skoularigis J, Louridas G, Butler J. The sympathetic nervous system in heart failure physiology, pathophysiology, and clinical implications. J Am Coll Cardiol. 2009 Nov 3;54(19):1747-62. doi: 10.1016/j.jacc.2009.05.015. PMID 19874988
- [Background] van de Port IG, Kwakkel G, Wittink H. Systematic review of cardiopulmonary exercise testing post stroke: Are we adhering to practice recommendations? J Rehabil Med. 2015 Nov;47(10):881-900. doi: 10.2340/16501977-2031. PMID 26551052
- [Background] Xiong L, Leung H, Chen XY, Han JH, Leung T, Soo Y, Wong E, Chan A, Lau A, Wong KS. Preliminary findings of the effects of autonomic dysfunction on functional outcome after acute ischemic stroke. Clin Neurol Neurosurg. 2012 May;114(4):316-20. doi: 10.1016/j.clineuro.2011.10.037. Epub 2011 Nov 15. PMID 22088362
- [Background] Vandermeeren Y, Jamart J, Ossemann M. Effect of tDCS with an extracephalic reference electrode on cardio-respiratory and autonomic functions. BMC Neurosci. 2010 Mar 16;11:38. doi: 10.1186/1471-2202-11-38. PMID 20233439
- See also: Related Info — http://stroke.ahajournals.org/content/early/2014/05/20/STR.0000000000000022
- See also: Related Info — http://dx.doi.org/10.1016/j.neubiorev.2016.05.001
- See also: Related Info — https://scholar.google.com.br/scholar?hl=pt-BR&q=Benef%C3%ADcios+da+fisioterapia+nas+sequelas+cr%C3%B4nicas+resultantes+de+acidente+vascular+encef%C3%A1lico+isqu%C3%AAmico+%E2%80%93+revis%C3%A3o+bibliogr%C3%A1fica&btnG=&lr=